CLINICAL TRIAL: NCT04026893
Title: Deceased Uterine Transplant in Absolute Uterine Infertility (AUIF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Stefan G Tullius, Chief, Division of Transplant Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001782/PHS
Record Dates: First submitted 2019-05-02; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Infertility of Uterine Origin
Keywords: AUFI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Uterine Transplant from Deceased Donor — The recipient will be started on anti-rejection medications (as is routine for transplant recipients) prior to the OR. Standard of care anesthesia and line placement will take place. The recipient will be appropriately identified as an organ recipient and the donor organ identified per required transplant protocols already in place. The recipient team will then connect the vasculature and appropriate supporting structures for the uterus transplant. Once the organ has been re-perfused, the remainder of the operation will take place and the patient will be moved to the Intensive Care Unit and later to the transplant patient floor for standard monitoring.

SUMMARY:
Our study will explore the feasibility of initiating a deceased donor uterine transplant program in addition to the existing living donor IRB at BWH.

Using the template established by teams around the world, we will identify emotionally and socially stable females of reproductive age with intact ovaries who are unable to gestate a child due to congenital or acquired uterine factor infertility. After careful screening, participants will undergo egg harvest, in vitro fertilization, and embryo cryopreservation using standard methods. Women who successfully complete the fertilization of at least six euploid embryos will be eligible to be placed on the waitlist for a deceased donor uterus transplant. After a successful transplant and a period of observation to ensure normal menstrual cycle and graft viability (anticipate six months), embryo implantation will be undertaken.

Following an embryo transfer, gestation will be carefully monitored by our high-risk pregnancy specialists. Medical research interventions include the surgical implantation of a uterus utilizing techniques by teams that have applied this approach successfully, close post-transplant follow up including immunosuppression therapy tailored to established standards during pregnancy minimizing fetal risks, and careful management of pregnancy. After childbearing is complete (at most two gestations), the donor uterus will be removed either during Cesarean or during an elective procedure. In addition, open ended interviews and surveys will be conducted to elicit ethical and psychosocial concerns arising from the experience of subjects and their families, health care providers, and the wider community. The investigator's intent is to monitor outcomes for transplant recipients as well as the live born infants for 30 days after removal of the transplanted uterus.

It is estimated that the time from screening to a potential live birth will be a minimum of 22 months, but likely between 24 - 36 months depending on organ availability.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of AUFI diagnosed by BWH gynecologist
* Ability to produce at least 6 euploid embryos for cryopreservation
* BMI ≤ 30
* GFR 60 or greater in any patient including those with a single kidney
* PRA 20% or less
* Deemed stable and capable of undergoing transplant by the transplant team to include psychiatry, social work, and transplant coordinator and study doctors to assure compliance with treatment
* Evidence to be compliant with follow-up and immunosuppression
* Partner willing to undergo psychological evaluation and receive immunizations as recommended
* Stable home environment to support a child

Exclusion Criteria:

* Active smoking, alcohol use or use of illicit drugs
* Inability to follow a strict medication dosing schedule post-transplant and adhere to required follow-up appointments.
* Any co-morbidities which would increase surgical risk, risk of pregnancy or the risk of taking anti-rejection medications as determined by the Maternal Fetal Specialist and Transplant Surgeon.
* Active infection: HIV, Hepatitis B, Hepatitis C
* Inadequate blood vessels to support the transplanted uterus.
* Prior extensive abdominal or pelvic surgery
* Presence of pelvic kidney
* History of abnormal PAP
* HPV related vulvar, vaginal or cervical dysplasia
* Evidence of genital condylomata
* History of PID
* One or more living biological children

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Live Births Following Uterus Transplant | Within 5 years of transplant
  To provide motherhood options for women with AUIF as an alternative to surrogacy or adoption, via gestating and giving birth via Cesarean section to a live infant.
Number of Surgically Successful Uterus Transplants | Within 3 months of transplant
  To achieve surgically successful uterus transplants.

SECONDARY OUTCOMES:
Financial impact of deceased donor uterus transplantation | Through Study completion, up to 5 years post transplant
  To analyze the overall impact of deceased donor uterus transplantation costs relative to established alternative procedures such as adoption and surrogacy.
Quality of life impact of deceased donor uterus transplantation | Through study completion, up to 5 years post transplant
  To analyze the overall impact of deceased donor uterus transplantation including changes in quality of life, relative to other established alternative procedures such as adoption and surrogacy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan G Tullius, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data will be published or presented at scientific meetings or distributed upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: For the duration of the study.
Access Criteria: Data will be published or presented at scientific meetings or distributed upon request.

REFERENCES:
- [Background] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Background] Tullius SG, Rudolf JA, Malek SK. Moving boundaries--the Nightingale twins and transplantation science. N Engl J Med. 2012 Apr 26;366(17):1564-5. doi: 10.1056/NEJMp1114193. No abstract available. PMID 22533575
- [Background] Lefkowitz A, Edwards M, Balayla J. The Montreal Criteria for the Ethical Feasibility of Uterine Transplantation. Transpl Int. 2012 Apr;25(4):439-47. doi: 10.1111/j.1432-2277.2012.01438.x. Epub 2012 Feb 23. PMID 22356169
- [Background] Del Priore G, Saso S, Meslin EM, Tzakis A, Brannstrom M, Clarke A, Vianna R, Sawyer R, Smith JR. Uterine transplantation--a real possibility? The Indianapolis consensus. Hum Reprod. 2013 Feb;28(2):288-91. doi: 10.1093/humrep/des406. Epub 2012 Nov 30. PMID 23202992
- [Background] McKay DB, Josephson MA. Pregnancy in recipients of solid organs--effects on mother and child. N Engl J Med. 2006 Mar 23;354(12):1281-93. doi: 10.1056/NEJMra050431. No abstract available. PMID 16554530